CLINICAL TRIAL: NCT00599417
Title: Prospective, Pivotal Unicentre, Randomized Double-bind, Placebo-controlled Study, to Evaluate Efficacy and Safety of Bacterial Lysates (Pulmonarom) in the Prevention of Respiratory Tract Infections
Brief Title: PulmonarOM (Bacterial Lysates) in Respiratory Tract Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BACLY_L_03329
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Bacterial Lysates

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Bacterial Lysates
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bacterial Lysates — Bacterial Lysates ampoules 3 mL, oral route, daily for 10 days, followed by 30 days free of medication and then 10 days of administration of the drug
  Arms: 1
Drug: placebo — placebo controlled
  Arms: 2

SUMMARY:
Primary

- To evaluate the efficacy of Pulmonaron in the decrease of interleukin-4/interferon gamma after second period of treatment

Secondary

* To evaluate the efficacy of Pulmonarom in the prevention of upper respiratory tract infections symptoms through patient evaluation of fever or respiratory presence after second period of treatment
* To evaluate loss of working or study days after second period of treatment
* To evaluate the safety and tolerability of Pulmonarom in the population under study

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of relapse or recurrence of respiratory infections or disease
* Patients with chronic respiratory disease as asthma, bronchitis or sinusitis

Exclusion Criteria:

* Patients unlikely to comply with the protocol, for example, uncooperativeness or impossibility to return for follow-up visits
* Patients who are participating or who have participated in another clinical trial during the previous 3 months
* Patients who have received immunology response stimulants during the previous 30 days
* Hypersensitivity

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Decrease of interleukin-4/interferon gamma index at baseline values | 60 days, 120 days

SECONDARY OUTCOMES:
Adverse events and laboratory evaluation | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Judith Diaz, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico